CLINICAL TRIAL: NCT01631812
Title: An Open-label Long-term Extension Trial From Late Phase II of SPM962 (243-05-001) in Advanced Parkinson's Disease Patients With Concomitant Treatment of L-dopa
Brief Title: A Long-Term Extension Trial From Late Phase II of SPM 962 in Advanced Parkinson's Disease Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Otsuka Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 243-06-001
Record Dates: First submitted 2012-06-25; First posted 2012-06-29 (Estimated); Results first posted 2014-03-19 (Estimated); Last update posted 2014-03-19 (Estimated); Status verified 2014-02

CONDITIONS: Parkinson's Disease
Keywords: SPM 962; rotigotine; Parkinson's disease; concomitant use of L-dopa
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SPM 962 (Experimental)
  Interventions: Drug: SPM 962

INTERVENTIONS:
Drug: SPM 962 — SPM 962 transdermal patch once a daily up to 36.0 mg/day

SUMMARY:
The primary objective of this study is to investigate safety of SPM 962 in advanced PD patients in a multi-center, open-label, non-controlled study following once-daily multiple transdermal doses of SPM962 within a range of 4.5 to 36.0 mg (maximum treatment period: 54 weeks). Efficacy is also to be exploratory investigated.

ELIGIBILITY:
Inclusion Criteria:

* Subject completed the preceding trial 243-05-001.

Exclusion Criteria:

* Subject discontinued from the preceding trial 243-05-001.
* Subject had a serious adverse event which association with the investigational drug was not ruled out during trial 243-05-001.
* Subject has a persistent serious adverse event at the baseline, which was observed and association with the investigational drug was ruled out during trial 243-05-001.
* Subject had persistent hallucination or delusion during trial 243-05-001.
* Subject has psychiatric conditions such as confusion, excitation, delirium, abnormal behaviour at the baseline.
* Subject has orthostatic hypotension at baseline.
* Subject has a history of epilepsy, convulsion etc. during trial 243-05-001.
* Subject has a complication of serious cardiac disorder.
* Subject has arrhythmia and need to be treated with class 1a antiarrhythmic drugs (e.g. quinidine, procainamide etc.) or class 3 antiarrhythmic drugs (e.g. amiodarone, sotalol etc.).
* Subject develops serious ECG abnormality at the baseline.
* Subject has QTc-interval >= 500 msec at the baseline or subject has an increase of QTc-interval >= 60 msec from the baseline in the trial 243-05-001 and has a QTc-interval > 470 msec in female or > 450 msec in male at the baseline.
* Subject had hypokalaemia in 243-05-001 study and not yet recovered.
* Subject has a total bilirubin >= 3.0 mg/dL or AST(GOT) or ALT(GPT) greater than 2.5 times of the upper limit of the reference range (or >= 100 IU/L) at the end of the period in trial 243-05-001.
* Subject has BUN >= 25 mg/dL or serum creatinine >= 2.0 mg/dl at the end of the taper period in trial 243-05-001.
* Subject has a history of allergic reaction to topical agents such as transdermal patch. Subject showed serious or extensive application site reactions beyond the application site in the 243-05-001 study.
* Subject who plans pregnancy during the trial.
* Subject has dementia.
* Subject is unable to give consent.
* Subject is judged to be inappropriate for this trial by the investigator for the reasons other than above.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2006-12; Primary Completion 2010-02 (Actual); Study Completion 2010-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyoji Imaoka, Mr, Study Director — Otsuka Pharmaceutical Co., Ltd.
Locations (7):
- Japan (7):
  - Chubu Region
  - Hokkaido Region
  - Kanto Region
  - Kinki Region
  - Kyushu Region
  - Shikoku Region
  - Tohoku Region

RESULTS

PARTICIPANT FLOW:
Groups:
- SPM 962: SPM 962 : SPM 962 transdermal patch once a daily up to 36.0 mg/day
Period: Overall Study
Arm/Group | SPM 962
Started | 130
Completed | 93
Not Completed | 37
Not completed — Adverse Event | 25
Not completed — Lack of Efficacy | 5
Not completed — Withdrawal by Subject | 4
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | SPM 962
Number analyzed (Participants) | 130
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 34
  >=65 years | 96
Age, Continuous [Mean (Standard Deviation); unit: years] | 66.9 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74
  Male | 56
Region of Enrollment [Number; unit: participants]
  Japan | 130

OUTCOME MEASURES:

1. Primary Outcome: Incidence and Severity of Adverse Events, Vital Signs, and Laboratory Parameters.
Description: Incidence and severity of adverse events, vital signs, and laboratory parameters after dosing.
  *decrease in difference between supine and standing systolic blood pressure
Time Frame: Up to 55 weeks after dosing
Population: Safety set (SS)
Measure: Number; unit: participants
Arm/Group | SPM 962
Number analyzed (Participants) | 130
participants
  Any AEs | 126
  Treatment-Related AEs | 112
  SAEs including death | 17
  Severe AEs | 12
  Discontinuation due to AEs | 26
  Severe laboratory abnormality | 10
  ≥30 mmHg decrease* | 6
  Treatment-related AE of orthostatic hypotension | 6
  QTcB ≥500 ms | 1

2. Secondary Outcome: Unified Parkinson's Disease Rating Scale (UPDRS) Part 3 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 3 sum score (on state) up to 54 weeks after dosing UPDRS is a scale for monitoring Parkinson's Disease-related disability and impairment. The UPDRS consists of the following four sub-scales. Part 1: Mentation, Part 2: Activities of Daily Living, Part 3: Motor, Part 4: Complications. Part 3 assesses 14 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, Up to 54 weeks after dosing
Population: Full analysis set (FAS), last observation carried forward (LOCF)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 129
Scores on a scale
  Week 12 | -9.6 (8.1)
  Week 24 | -9.1 (8.2)
  Week 52 | -8.3 (9.8)

3. Secondary Outcome: UPDRS Part 2 Sum Score
Description: Mean change (LOCF) from baseline in UPDRS Part 2 sum score (average scores of on state and off state) up to 54 weeks after dosing UPDRS sub-scale Part 2 assesses 13 items. Each item is scored from 0 (normal) to 4 (severe). The sum score serves as the sub-scale score. A higher score indicates a greater severity of symptoms. Thus a decrease in the scores means improvement.
Time Frame: Baseline, Up to 54 weeks after dosing
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | SPM 962
Number analyzed (Participants) | 129
Scores on a scale
  Week 12 | -2.7 (3.5)
  Week 24 | -2.4 (3.7)
  Week 52 | -1.9 (4.7)

4. Secondary Outcome: Absolute Time Spent "Off"
Description: Mean number of hours in "off state" during a 24-hour period.
Time Frame: Up to 54 weeks after dosing
Population: FAS subjects with "off state" at baseline
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | SPM 962
Number analyzed (Participants) | 84
Hours
  Week 12 | -3.0 (2.7)
  Week 24 | -2.6 (2.9)
  Week 52 | -1.9 (3.0)

5. Primary Outcome: Skin Irritation Score of the Application Site
Description: Skin irritation score of the application site were evaluated according to the criteria below. The worst score throughout the treatment period was used in the analysis.
  -: no reaction, ±: mild erythema, +: erythema, ++: erythema and Oedema, +++: erythema and oedema and rash papular, or serous papule, or vesicles, ++++: bullosum
Time Frame: Up to 55 weeks after dosing
Population: SS
Measure: Number; unit: participants
Arm/Group | SPM 962
Number analyzed (Participants) | 130
participants
  - | 18
  ± | 53
  + | 42
  ++ | 9
  +++ | 7
  ++++ | 1
  +++> | 8

ADVERSE EVENTS:
Time Frame: 54 weeks
Arm/Group | SPM 962
Serious Adverse Events (participants affected / at risk) | 17/130
Other Adverse Events (participants affected / at risk) | 119/130
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM 962 (N=130)
Colonic Polyp (Gastrointestinal disorders) | 1 (1)
Sudden Death (General disorders) | 1 (1)
Bile Duct Stone (Hepatobiliary disorders) | 1 (1)
Atypical Mycobacterial Infection (Infections and infestations) | 1 (1)
Herpes Zoster (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 2 (2)
Pelvic Fracture (Injury, poisoning and procedural complications) | 1 (1)
Weight Decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Diabetes Mellitus (Metabolism and nutrition disorders) | 1 (1)
Rheumatoid Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Carcinoma Kidney (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large Intestine Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Delusion (Psychiatric disorders) | 2 (2)
Hallucination (Psychiatric disorders) | 1 (1)
Hallucination, Auditory (Psychiatric disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | SPM 962 (N=130)
Anaemia (Blood and lymphatic system disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 17 (24)
Constipation (Gastrointestinal disorders) | 13 (13)
Vomiting (Gastrointestinal disorders) | 11 (13)
Diarrhoea (Gastrointestinal disorders) | 6 (6)
Toothache (Gastrointestinal disorders) | 4 (5)
Application Site Reaction (General disorders) | 67 (69)
Oedema Peripheral (General disorders) | 8 (8)
Application Site Erythema (General disorders) | 4 (5)
Feeling Abnormal (General disorders) | 4 (5)
Nasopharyngitis (Infections and infestations) | 27 (37)
Cystitis (Infections and infestations) | 4 (4)
Tinea Infection (Infections and infestations) | 4 (4)
Contusion (Injury, poisoning and procedural complications) | 15 (19)
Fall (Injury, poisoning and procedural complications) | 10 (14)
Excoriation (Injury, poisoning and procedural complications) | 4 (4)
Tooth Fracture (Injury, poisoning and procedural complications) | 4 (4)
Blood Creatine Phosphokinase Increased (Investigations) | 8 (11)
Weight Decreased (Investigations) | 5 (5)
Decreased Appetite (Metabolism and nutrition disorders) | 4 (5)
Back Pain (Musculoskeletal and connective tissue disorders) | 13 (16)
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 (5)
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 4 (4)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 4 (4)
Dyskinesia (Nervous system disorders) | 21 (24)
Dizziness (Nervous system disorders) | 10 (13)
Headache (Nervous system disorders) | 7 (7)
Dystonia (Nervous system disorders) | 5 (6)
Dizziness Postural (Nervous system disorders) | 4 (6)
Hallucination Visual (Psychiatric disorders) | 20 (28)
Somnolence (Psychiatric disorders) | 19 (20)
Insomnia (Psychiatric disorders) | 8 (8)
Hallucination (Psychiatric disorders) | 5 (5)
Upper Respiratory Tract Inflammation (Respiratory, thoracic and mediastinal disorders) | 10 (12)
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Eczema (Skin and subcutaneous tissue disorders) | 4 (4)
Rash (Skin and subcutaneous tissue disorders) | 4 (5)
Orthostatic Hypotension (Vascular disorders) | 7 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No